CLINICAL TRIAL: NCT01391559
Title: Efficacy of Inhaling Bronchodilator Medications in Patients With Chronic Obstructive Pulmonary Disease Who Have a Low Peak Inspiratory Flow Rate
Brief Title: Efficacy of Inhaling Bronchodilator Medications in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CPHS22812
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: breathing difficulty
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Formoterol Fumarate; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arformoterol (Experimental): beta-2 agonist bronchodilator
  Interventions: Drug: arformoterol
- salmeterol (Active Comparator): beta-2 agonist bronchodilator
  Interventions: Drug: salmeterol

INTERVENTIONS:
Drug: arformoterol — 15 mcg administered via nebulizer
  Other Names: Brovana
  Arms: arformoterol
Drug: salmeterol — 50 mcg delivered vis Diskus
  Other Names: Serevent
  Arms: salmeterol

SUMMARY:
Some patients with Chronic Obstructive Pulmonary Disease (COPD) report that they are uncertain whether they achieve clinical benefit using a dry-powder inhaler (DPI). One possible explanation is that the patient is unable to inhale the dry powder bronchodilator medication into the lower respiratory tract due to a low peak inspiratory flow rate (PIFR). A PIFR < 60 l/min is considered to be suboptimal flow for a DPI, including the Diskus device. The hypothesis of the study is that the forced expiratory volume in 1 second (FEV1) measured at two hours after inhalation of the study medication will be higher with arformoterol solution (15 mcg) from a nebulizer compared with salmeterol dry powder (50 mcg) inhaled from the Diskus.

ELIGIBILITY:
Inclusion Criteria:

* male or female patient 60 years of age or older; diagnosis of COPD; current or former smoker; previous or current use of Diskus device; PIFR < 60 l/min using the In-check DIAL against the resistance of the Diskus device; clinically stable.

Exclusion Criteria:

* any patient who has a concomitant disease that might interfere with study procedures or evaluation; inability to withhold short-acting and long-acting bronchodilators on the days of testing

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald A Mahler, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] Janssens W, VandenBrande P, Hardeman E, De Langhe E, Philps T, Troosters T, Decramer M. Inspiratory flow rates at different levels of resistance in elderly COPD patients. Eur Respir J. 2008 Jan;31(1):78-83. doi: 10.1183/09031936.00024807. Epub 2007 Sep 26. PMID 17898020
- [Derived] Mahler DA, Waterman LA, Ward J, Gifford AH. Comparison of dry powder versus nebulized beta-agonist in patients with COPD who have suboptimal peak inspiratory flow rate. J Aerosol Med Pulm Drug Deliv. 2014 Apr;27(2):103-9. doi: 10.1089/jamp.2013.1038. Epub 2013 Jun 8. PMID 23745526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: July 2011 to October 2012; Location: medical clinic
Pre-assignment Details: 26 patients screened: 5 excluded because did not meet exclusion criteria; 1 excluded because of exacerbation after visit 1.
Groups:
- Arformoterol First, Then Salmeterol: Arformoterol (15 mcg/2 mL) solution via nebulizer in the first intervention, Salmeterol (50 mcg) Diskus in the second intervention
- Salmeterol First, Then Arformoterol: Salmeterol (50 mcg) Diskus in the first intervention, Arformoterol (15 mcg/2 mL) solution via nebulizer in the second intervention
Period: First Intervention
Arm/Group | Arformoterol First, Then Salmeterol | Salmeterol First, Then Arformoterol
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Arformoterol First, Then Salmeterol | Salmeterol First, Then Arformoterol
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive Arformoterol first and Salmeterol first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 71 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1) From Baseline at Two Hours After Inhalation of the Study Medication
Description: FEV1
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Arformoterol: Arformoterol aerosol solution (15 mcg/2 mL)via nebulizer
- Salmeterol: Salmeterol dry powder (50 mcg) via Diskus
Arm/Group | Arformoterol | Salmeterol
Number analyzed (Participants) | 10 | 10
mL | 84 (72) | 52 (105)
Statistical Analysis 1: Comparison: Arformoterol vs Salmeterol; Test type: Superiority or Other; p = 0.17, t-test, 2 sided; Mean Difference (Final Values) = 32

ADVERSE EVENTS:
Arm/Group | Arformoterol | Salmeterol
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No